CLINICAL TRIAL: NCT01409694
Title: Evaluation d'Une stratégie thérapeutique d'Association médicamenteuse Pour la Prise en Charge de la Maladie d'Alzheimer et Des Maladies apparentées au Stade modéré
Brief Title: Alzheimer's Disease - Input of Vitamin D With mEmantine Assay
Acronym: AD-IDEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-024506-35
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Vitamin D; Cholecalciferol; Memantine; Cognition Disorders
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders | interventions — Memantine; Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): All participants start the treatment with memantine on the first day of the study and immediately start vitamin D supplementation.
  Interventions: Drug: Memantine; Drug: Vitamin D
- Placebo (Placebo Comparator): Participants in this arm start the treatment with memantine in the same way as the 'Intervention' group. They also immediately start Vitamin D placebo administered at the same pace.
  Interventions: Drug: Memantine; Drug: Vitamin D placebo

INTERVENTIONS:
Drug: Memantine — Memantine is administered to all participants according to the usual strategy, with upward titration of 5 mg per week during the first three weeks to reduce the risk of side effects. The final dosage is 20 mg per day, with no subsequent modification of dosage or specialty during the trial.
  Other Names: Chlorhydrate de mémantine (Ebixa®)
Drug: Vitamin D — Subjects receive Vitamin D supplementation (cholecalciferol 100,000 IU, drinking solution, 2 mL vial) at a rate of 1 drinking vial of 100,000 IU cholecalciferol every month. In brief, the total dose is 600,000 IU over the duration of the study starting with one vial at the time of inclusion, then at week(W) 4, W8, W12, W16 and W20. The dose of vitamin D supplementation will not be adjusted except in case of an adverse event such as hypercalcemia. In this case, vitamin D supplementation is stopped and the participant is released prematurely from the study.
  Other Names: Colecalciferol
  Arms: Intervention
Drug: Vitamin D placebo — Subjects receive Vitamin D placebo (drinking solution, 2mL vial) at a rate of 1 drinking vial every month. In brief, the subjects start with one vial at the time of inclusion, then at week(W)4, W8, W12, W16 and W20. The placebo drinking solution contains all the excipients present in the Vitamin D vial.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect after 24 weeks of the oral intake of vitamin D3 (cholecalciferol) with the effect of a placebo on the change of cognitive performance in patients suffering from moderate Alzheimer's disease or related disorders (ADRD) and receiving memantine.

DETAILED DESCRIPTION:
Current treatments for Alzheimer's disease and related disorders (ADRD) are symptomatic and can only temporarily slow down ADRD. Future possibilities of care could rely on multi-target drugs therapies that address simultaneously several pathophysiological processes leading to neurodegeneration. We hypothesized that the combination of memantine with vitamin D could be neuroprotective in ADRD, thereby limiting neuronal loss and cognitive decline.

The primary objective of this trial is to compare the effect after 24 weeks of the oral intake of vitamin D3 with the effect of a placebo on the evolution of cognitive performance in patients suffering from moderate ADRD and receiving memantine.

The secondary objectives of the study are as follows:

* To compare the effect after 12 weeks of the oral intake of vitamin D3 with the effect of a placebo on the evolution of cognitive performance in patients suffering from moderate ADRD and receiving memantine.
* To compare the effect after 12 and 24 weeks of the oral intake of vitamin D3 with the effect of a placebo on the evolution of functional abilities in patients suffering from moderate ADRD and receiving memantine.
* To compare the effect after 12 and 24 weeks of the oral intake of vitamin D3 with the effect of a placebo on the evolution of postural and gait performance in patients suffering from moderate ADRD and receiving memantine.
* To determine the compliance to treatment and tolerance of the oral intake of vitamin D3 in patients suffering from moderate ADRD and receiving memantine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Diagnosis of moderate Alzheimer's disease or related disorders (DSM-IV/NINCDSADRDA) with a score of Mini-Mental State Examination (MMSE) between 10 and 20 inclusively
* To have hypovitaminosis D (i.e., serum 25-hydroxyvitamin D [25OHD]concentration < 30 ng/mL)
* To have no hypercalcemia (defined as serum calcium concentration ≥ 2,65 mmol/L)
* To have given and signed an informed consent form to participate in the trial (or informed consent form obtained from the trusted person or legal representative, as appropriate)
* To be affiliated to French Social Security

Exclusion Criteria:

* The use of standard antidementia drugs (i.e., anticholinesterasics, memantine, or vasodilatators) in the past 60 days
* Severe hepatic or renal failure
* Severe, unstable or poorly controlled medical conditions at the time of the inclusion
* Other cognitive disorders (untreated dysthyroid, deficiency in vitamin B9 or B12, chronic ongoing ethylism, history of syphilis, stroke, delirium revealed with the Confusion Assessment Method (CAM), severe depressive symptomatology (Geriatric Depression score ≥ 10/15))
* Contra-indications to memantine or vitamin D
* Enrollment in another simultaneous clinical trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  Cognitive performance is measured with Alzheimer's Disease Assessment Scale-cognition score (ADAS-cog)

SECONDARY OUTCOMES:
Change in other cognitive scores | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  MMSE, Cognitive Assessment Battery, Frontal Assessment Battery, Trail Making Test parts A and B
Change in functional performance | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  Activities of Daily Living scale and 4-item Instrumental Activities of Daily Living scale
Change in posture and gait | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  Timed Up & Go, Five Time Sit-to-Stand and spatio-temporal analysis of walking
Between-group comparison of compliance to treatment and tolerance | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  These outcomes are assessed together with the serum concentrations of 25OHD, calcium and parathyroid hormone.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Annweiler, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Annweiler C, Beauchet O. Possibility of a new anti-alzheimer's disease pharmaceutical composition combining memantine and vitamin D. Drugs Aging. 2012 Feb 1;29(2):81-91. doi: 10.2165/11597550-000000000-00000. PMID 22233455
- [Derived] Annweiler C, Fantino B, Parot-Schinkel E, Thiery S, Gautier J, Beauchet O. Alzheimer's disease--input of vitamin D with mEmantine assay (AD-IDEA trial): study protocol for a randomized controlled trial. Trials. 2011 Oct 20;12:230. doi: 10.1186/1745-6215-12-230. PMID 22014101